CLINICAL TRIAL: NCT02955355
Title: Long-Term Tolerability and Safety of Immune Globulin Infusion 10% (Human) With Recombinant Human Hyaluronidase (HYQVIA/HyQvia) for the Treatment of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Long-Term Tolerability and Safety of HYQVIA/HyQvia in CIDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 161505; 2016-000374-37 (EudraCT Number)
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HYQVIA/HyQvia (Experimental): Participants received HYQVIA/HyQvia (recombinant human hyaluronidase [rHuPH20] at a dose of 80 units per gram (U/g) immunoglobulin G [IgG], followed by subcutaneous [SC] immune globulin infusion [IGI] 10%) at the same monthly equivalent dose as the individual participant's IgG treatment in Study 161403, every 3 or 4 weeks in this Extension Study for 77.3 months or until relapse.
  Interventions: Biological: HYQVIA

INTERVENTIONS:
Biological: HYQVIA — Participants received HYQVIA/HyQvia SC which contains both Immune Globulin Infusion 10% (Human) (IGI, 10%) and recombinant human hyaluronidase (rHuPH20).
  Other Names: 10%) with recombinant human hyaluronidase (rHuPH20); Immune Globulin Infusion 10% (Human) (IGI; IGI

SUMMARY:
Adults with Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) who have completed study 161403 will be able to take part in this study.

The main aim of the study is to evaluate side effects in the long-term treatment with HYQVIA/HyQvia.

All participants will receive HYQVIA/HyQvia in the same way as they were receiving in study 161403. The dosing interval of HYQVIA/HyQvia can be adjusted after 12 weeks of treatment in study 161505 if the study doctor determines that it is safe to do so.

Participants will visit the clinic within 1 week after the first and second dose of HYQVIA/HyQvia and then every 12 weeks for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Has completed Epoch 1 of Study 161403 without CIDP worsening.
2. If female of childbearing potential, the participant must have a negative pregnancy test at baseline and agree to employ adequate birth control measures (eg, birth control pills/patches, intrauterine device, or diaphragm or condom [for male partner] with spermicidal jelly or foam) throughout the course of the study.

Exclusion Criteria:

1. Participant has a serious medical condition such that the participant's safety or medical care would be impacted by participation in this Extension Study.
2. New medical condition that developed during participation in study 161403 that, in the judgment of the investigator, could increase risk to the participant or interfere with the evaluation of investigational medicinal product (IMP) and/or conduct of the study.
3. Participant is scheduled to participate in another non-Baxalta clinical study involving an IP or investigational device during the course of this study.
4. The participant is nursing or intends to begin nursing during the course of the study
5. Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study (with the exception of study 161403) involving an IP or investigational device during the course of this study.
6. The participant is a family member or employee of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (35):
- Arizona Neuromuscular Research Center, Phoenix, Arizona, United States
- Hosp.Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires, Argentina
- Instituto de Neurologia de Curitiba - Hospital Ecoville, Curitiba, Paraná, Brazil
- Canada (3):
  - University of Alberta Hospital, Edmonton, Alberta
  - LHSC - University Hospital, London, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
- Institucion Prestadora de Servicios de Salud de la Universidad de Antioquia "IPS UNIVERSITARIA", Medellín, Colombia
- Czechia (2):
  - Fakultni nemocnice Ostrava, Ostrava, Poruba
  - Fakultni nemocnice v Motole, Prague
- Århus Universitetshospital, Aarhus C, Denmark
- France (3):
  - CHU de Nice, Nice, Alpes Maritimes
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - Hopital Neurologique Pierre Wertheimer, Bron, Rhone
- Universitaetsklinikum Leipzig AoeR, Leipzig, Saxony, Germany
- University Hospital of Patra, Pátrai, Greece
- Italy (5):
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine
- Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City, Mexico
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Nis, Niš
- Fakultna nemocnica Nitra, Nitra, Slovakia
- Hospital Universitari Vall d'Hebron, Barcelona, Spain
- Turkey (Türkiye) (4):
  - Pamukkale Uni. Med. Fac., Denizli
  - Dokuz Eylul University Faculty of Medicine, Izmir
  - Selcuk Universitesi Selcuklu Tip Fakultesi Hastanesi, Konya
  - Celal Bayar University Medical Faculty, Manisa
- United Kingdom (2):
  - King's College Hospital, London, Greater London
  - The Walton Centre, Liverpool, Merseyside

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45c9a

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 39 investigative sites worldwide from 14 November 2016 to 04 July 2023.
Pre-assignment Details: A total of 85 participants with a diagnosis of chronic inflammatory demyelinating polyradiculoneuropathy (CIDP) who completed Study 161403 (NCT02549170) without CIDP worsening were enrolled in this Extension Study to receive HYQVIA/HyQvia.
Period: Overall Study
Arm/Group | HYQVIA/HyQvia
Started | 85
Completed | 0
Not Completed | 85
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Physician Decision | 21
Not completed — Site Terminated by Sponsor | 35
Not completed — Withdrawal by Subject | 19
Not completed — Reason Not Specified | 5

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication.
Groups:
- HYQVIA/HyQvia: Participants received HYQVIA/HyQvia (rHuPH20 at a dose of 80 U/g IgG, followed by SC IGI 10%) at the same monthly equivalent dose as the individual participant's IgG treatment in Study 161403, every 3 or 4 weeks in this Extension Study for 77.3 months or until relapse.
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (13.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 81
  More than one race | 0
  Unknown or Not Reported | 3
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 171.5 (10.98)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 80.89 (18.856)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter square (kg/m^2)] — BMI = weight (kg)/[height (m)^2]
  kilograms per meter square (kg/m^2) | 27.42 (5.587)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Serious Adverse Events (SAEs) and Adverse Events (AEs), Regardless of Causality
Description: An AE was defined as any untoward medical occurrence in a participant administered an investigational product (IP) that did not necessarily have a causal relationship with the treatment. An SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death, was life-threatening, required inpatient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. Treatment emergent adverse events (TEAEs) were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants
  Any TEAE | 76
  Any Serious TEAE | 20

2. Primary Outcome: Number of Participants With Causally Related Treatment-emergent SAEs and AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. An SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death, was life-threatening, required inpatient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Causality was used to determine whether there was a reasonable possibility that the IP was etiologically related to/associated with the AE.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants
  Any IP-Related TEAE | 51
  Any IP-Related Serious TEAE | 3

3. Primary Outcome: Number of Participants With Adverse Reactions (ARs) or Suspected Adverse Reactions (SARs) Categorized as Serious and Non-serious
Description: An AR plus SAR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 hours following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Serious AR/SAR=any AR/SAR that is an untoward medical occurrence which at any dose meets one or more of following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of existing hospitalization, results in persistent or significant disability/incapacity,is a congenital anomaly/birth defect,is a medically important event,thromboembolic events,hemolytic anemia. Nonserious AR/SAR=AR/SAR that does not meet the criteria.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants
  Any Serious AR/SAR | 7
  Any Non-serious AR/SAR | 57

4. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events That May be a Result of Immune-Mediated Responses
Description: Percentage of participants with TEAEs that may be a result of immune-mediated response to either immunoglobulin, rHuPH20, or other factors such as allergic reactions, immune complex-mediated reactions: local, complex-mediated reactions: systemic, thrombotic and embolic events were assessed. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. The percentage was rounded off to the nearest decimal.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
percentage of participants | 7.1

5. Primary Outcome: Number of Treatment-Emergent SAEs and AEs Associated With Infusions, Regardless of Causality
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. An SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death, was life-threatening, required inpatient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. AEs associated with an infusion are defined as AEs occurring after administration of IP (or any TEAE). Participants can have more than one TEAE associated with infusion.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: events in participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
events in participants
  Serious TEAEs | 30
  TEAEs | 1406

6. Primary Outcome: Number of Causally Related Treatment-Emergent SAEs and AEs Associated With Infusions
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. An SAE was defined as an untoward medical occurrence that at any dose met one or more of the following criteria: outcome was fatal/resulted in death, was life-threatening, required inpatient hospitalization or resulted in prolongation of an existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. AEs associated with an infusion are defined as AEs occurring after administration of IP (or any TEAE). Causality was used to determine whether there was a reasonable possibility that the IP was etiologically related to/associated with the AE.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: events in participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
events in participants
  IP-Related Serious TEAEs | 3
  IP-Related TEAEs | 798

7. Primary Outcome: Number of TEAEs Temporally Associated With Infusions
Description: TEAEs that occurred during infusion or within 72 hours post-infusion were considered to be temporally associated with infusions. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Participants can have more than one TEAE temporally associated with infusion.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: events in participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
events in participants | 857

8. Primary Outcome: Number of Serious and Non-Serious ARs or SARs Associated With Infusions
Description: An AR/SAR=any AE that meets any of following criteria: AE considered by either investigator and/or sponsor to be possibly or probably related to IP administration, begins during infusion of IP or within 72 hours following end of IP infusion,or AE for which causality assessment is missing or indeterminate. ARs/SARs associated with an infusion=AEs considered by the investigator to be occurring after administration of IP. Serious AR/SAR=any AR/SAR that is an untoward medical occurrence which at any dose meets one or more of following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of existing hospitalization, results in persistent or significant disability/incapacity,is a congenital anomaly/birth defect,is a medically important event,thromboembolic events,hemolytic anemia. Nonserious AR/SAR=AR/SAR that does not meet the criteria. Participants can have more than one AR/SAR associated with infusion.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: events in participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
events in participants
  Serious ARs/SARs | 8
  Non-Serious ARs/SARs | 913

9. Primary Outcome: Number of Infusions Associated With One or More Systemic TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the Medical Dictionary for Regulatory Activities (MedDRA) Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Infusions associated with one or more AEs are defined as follows: if an AE occurs after an infusion but prior to the next infusion that infusion is associated with that AE.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: infusions
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
infusions | 50

10. Primary Outcome: Number of Infusions Associated With One or More Local TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Infusions associated with one or more AEs are defined as follows: if an AE occurs after an infusion but prior to the next infusion that infusion is associated with that AE.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: infusions
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
infusions | 17

11. Primary Outcome: Number of Infusions for Which the Infusion Rate Was Reduced and/or the Infusion Was Interrupted or Stopped Due to Intolerability and/or TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: infusions
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
infusions | 3

12. Primary Outcome: Rate of TEAEs Categorized as Systemic and Local Regardless of Causality, Expressed as Number of Events Per Infusion
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Data for number of events per infusion was assessed at the group level calculated by dividing number of events by total number of infusions administered to participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/infusion
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
AEs/infusion
  Systemic TEAEs | 0.25
  Local TEAEs | 0.15

13. Primary Outcome: Rate of TEAEs Categorized as Systemic and Local Regardless of Causality, Expressed as Number of Events Per Participant
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Data for number of events per participant was assessed at the group level calculated by dividing number of events by total number of participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/participant
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
AEs/participant
  Systemic TEAEs | 10.38
  Local TEAEs | 6.16

14. Primary Outcome: Rate of TEAEs Categorized as Systemic and Local Regardless of Causality, Expressed as Number of Events Per 1000 Participant-year
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Events per participant-years was calculated as follows: 1000 x (number of events / total number of days of exposure, i.e., the sum of duration of treatment for all participants in the Safety Analysis Set, divided by 365.25).
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/1000 participant-year
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
AEs/1000 participant-year
  Systemic TEAEs | 4000.23
  Local TEAEs | 2376.55

15. Primary Outcome: Rate of IP-Related TEAEs Categorized as Systemic and Local, Expressed as Number of Events Per Infusion
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". An adverse event that was "possibly related" or "probably related" to IP, or for which the relationship was unknown or missing, was considered as a "related AE". Data for number of events per infusion was assessed at the group level calculated by dividing number of events by total number of infusions administered to participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/infusion
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
AEs/infusion
  Systemic IP-Related TEAEs | 0.08
  Local IP-Related TEAEs | 0.15

16. Primary Outcome: Rate of IP-Related TEAEs Categorized as Systemic and Local, Expressed as Number of Events Per Participant
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". An adverse event that was "possibly related" or "probably related" to IP, or for which the relationship was unknown or missing, was considered as a "related AE". Data for number of events per participant was assessed at the group level calculated by dividing number of events by total number of participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/participant
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
AEs/participant
  Systemic IP-Related TEAEs | 3.38
  Local IP-Related TEAEs | 6.01

17. Primary Outcome: Rate of IP-Related TEAEs Categorized as Systemic and Local, Expressed as Number of Events Per 1000 Participant-year
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. Systemic TEAEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local TEAEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". An adverse event that was "possibly related" or "probably related" to IP, or for which the relationship was unknown or missing, was considered as a "related AE". Events per participant-years was calculated as follows: 1000 x (number of events / total number of days of exposure, i.e., the sum of duration of treatment for all participants in the Safety Analysis Set, divided by 365.25).
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/1000 participant-year
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
AEs/1000 participant-year
  Systemic IP-Related TEAEs | 1301.66
  Local IP-Related TEAEs | 2317.59

18. Primary Outcome: Rate of ARs or SARs Categorized as Local and Systemic, Expressed as Reactions Per Infusion
Description: An AR plus SAR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 hours following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Systemic AEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local AEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Data for number of events per infusion was assessed at the group level calculated by dividing number of events by total number of infusions administered to participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: reactions/infusion
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
reactions/infusion
  Systemic ARs/SARs | 0.11
  Local ARs/SARs | 0.15

19. Primary Outcome: Rate of ARs or SARs Categorized as Local and Systemic, Expressed as Reactions Per Participant
Description: An AR plus SAR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 hours following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Systemic AEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local AEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Data for number of events per participant was assessed at the group level calculated by dividing number of events by total number of participants in the Safety Analysis Set.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: reactions/participant
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
reactions/participant
  Systemic ARs/SARs | 4.58
  Local ARs/SARs | 6.16

20. Primary Outcome: Rate of ARs or SARs Categorized as Local and Systemic, Expressed as Reactions Per 1000 Participant-year
Description: An AR plus SAR is any AE that meets any of the following criteria: an AE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or that begins during infusion of IP or within 72 hours following the end of IP infusion, or AE for which causality assessment is missing or indeterminate. Systemic AEs were defined as AEs that were not included in the MedDRA Higher Level Group Term "administration site reactions" and did not contain the phrase "injection site". Local AEs were defined as AEs that were included in the MedDRA Higher Level Group Term "administration site reactions" or contained the phrase "injection site" or "infection site". Events per participant-years was calculated as follows: 1000 x (number of events / total number of days of exposure, i.e., the sum of duration of treatment for all participants in the Safety Analysis Set, divided by 365.25).
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: reactions/1000 participant-year
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
reactions/1000 participant-year
  Systemic ARs/SARs | 1764.27
  Local ARs/SARs | 2376.55

21. Primary Outcome: Number of Participants With a TEAE That Led to Discontinuation From Study
Description: as for outcome 11
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants | 4

22. Primary Outcome: Number of Participants With Moderate or Severe TEAEs That May be a Result of Immune-Mediated Responses
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. A moderate or severe AE could be a result of immune-mediated response to either immunoglobulin, rHuPH20, or other factors such as allergic reactions, immune complex-mediated reactions: local, complex-mediated reactions: systemic, thrombotic and embolic events. The severity of each AE was assessed by the investigator using clinical expertise based on the following description: moderate=AE produces limited impairment of function and may require therapeutic intervention and produces no sequela/sequelae; severe=AE results in a marked impairment of function and may lead to temporary inability to resume usual life pattern and produces sequela/sequelae, which require (prolonged) therapeutic intervention.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants | 3

23. Primary Outcome: Rate of Moderate or Severe TEAEs That May be a Result of Immune-Mediated Responses, Expressed as Number of Events Per 100 Infusions
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that did not necessarily have a causal relationship with the treatment. TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. A moderate or severe AE could be a result of immune-mediated response to either immunoglobulin, rHuPH20, or other concomitant medications. The severity of each AE was assessed by the investigator using clinical expertise. Data for number of events per 100 infusions was assessed at the group level calculated by dividing number of events by total number of infusions and multiplying that by 100.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Number; unit: AEs/100 infusions
Units Other Than Participants: infusions
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Number analyzed (infusions) | 3487
AEs/100 infusions | 0.0860

24. Primary Outcome: Number of Participants That Experienced Treatment-Emergent Local Infusion Site Reactions
Description: TEAEs were defined as adverse events that occurred during or after administration of the first dose of IP in this Extension Study. AE=any untoward medical occurrence in participant administered an IP that does not have causal relationship with treatment. Adverse reaction/suspected adverse reaction=AE that is considered by the investigator to be possibly or probably related to IP administration, or for which the causality is indeterminate or missing, or that begins during infusion of IP or within 72 hours following the end of IP infusion. All local infusion site treatment-emergent AEs were reported as adverse reactions.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants | 30

25. Primary Outcome: Number of Participants With Treatment-Emergent Local Tolerability Events During Ramp-up
Description: Participants with local tolerability events were those for which the infusion rate was reduced and/or the infusion was interrupted or stopped due to intolerability and/or AEs. These events were assessed during the initial ramp-up for each participant i.e., during the first 8 weeks of open-label extension study 161505 [NCT02955355] among participants originally randomized to placebo (as being in the placebo arm, they had no ramp-up during the 161403 [NCT02549170] study) versus during the 8-week ramp-up for participants originally randomized to active HYQVIA in double-blind 161403 study. Thus, the data for this outcome measure are presented per the bifurcation of participants in the study 161403.
Time Frame: During the ramp-up (8 weeks)
Population: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication. As prespecified in the statistical analysis plan (SAP), comparative local tolerability data for the ramp-up of 8 weeks from studies 161403 (for participants originally randomized to HYQVIA in double-blind) and 161505 were reported in the results of study 161505.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Then HYQVIA/HyQvia: Participants received placebo in the study 161403 and received HYQVIA/HyQvia (rHuPH20 at a dose of 80 U/g IgG, followed by SC IGI 10%) at the same monthly equivalent dose as the individual participant's IgG treatment in Study 161403, every 3 or 4 weeks in this Extension Study for 77.3 months or until relapse.
- HYQVIA/HyQvia Then HYQVIA/HyQvia: Participants received HYQVIA/HyQvia in the study 161403 and received HYQVIA/HyQvia (rHuPH20 at a dose of 80 U/g IgG, followed by SC IGI 10%) at the same monthly equivalent dose as the individual participant's IgG treatment in Study 161403, every 3 or 4 weeks in this Extension Study for 77.3 months or until relapse.
Arm/Group | Placebo Then HYQVIA/HyQvia | HYQVIA/HyQvia Then HYQVIA/HyQvia
Number analyzed (Participants) | 42 | 43
Participants | 6 | 13

26. Primary Outcome: Number of Participants With Local Infusion Reactions, as a Function of Dosing Interval, Infusion Rate Per Site, and Infusion Volume Per Site
Description: Local infusion reactions were defined as local (administration site-related) adverse events. Median infusion rate per site was derived as the median value across all participants, per participant's average infusion rate, by site: actual volume infused / duration in hours of infusion / number of sites. Median infusion volume per site was derived as the median value across all participants, per participant's average actual volume infused, by site: actual volume infused / number of sites. Number of participants with local infusion reactions as a function of each of the categories are presented below.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication. Overall number analyzed is the number of participants with local infusion reactions.
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 30
Participants
  3 Week Dosing Interval | 8
  4 Week Dosing Interval | 22
  < Median Infusion Rate per Site | 15
  ≥ Median Infusion Rate per Site | 15
  < Median Infusion Volume per Site | 15
  ≥ Median Infusion Volume per Site | 15

27. Primary Outcome: Number of Participants Whose Anti-Hyaluronidase Binding Antibody Titers Rose by ≥4-fold From Baseline
Description: Number of participants whose anti-hyaluronidase antibody titers rose by ≥4 fold from the baseline value at any point during the study was assessed.
Time Frame: Baseline, up to 6.6 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants | 16

28. Primary Outcome: Number of Participants With Binding Antibodies to rHuPH20
Description: Binding antibodies were defined as anti-rHuPH20 titer ≥1:160.
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication. Overall number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 84
Participants | 14

29. Primary Outcome: Number of Participants With Neutralizing Antibodies Binding to rHuPH20
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 84
Participants | 2

30. Primary Outcome: Number of Participants With a Decline of Anti-rHuPH20 Binding Antibody Titers to the Antibody Titer Level at Baseline in Study 161403 or to <1:160 Antibody Titer Level at the Study Completion or Early Discontinuation
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 85
Participants | 12

31. Primary Outcome: Number of Participants Who Had >1:10,000 Anti-rHuPH20 Binding Antibody Titers With Neutralizing Antibodies
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication. Overall number analyzed is the number of participants who had >1:10,000 anti-rHuPH20 antibody titers.
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 8
Participants | 2

32. Secondary Outcome: Number of Participants Who Had >1:10,000 Anti-rHuPH20 Binding Antibody Titers Showing Cross Reactivity With Hyaluronidase (Hyal)-1,2 and 4
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | HYQVIA/HyQvia
Number analyzed (Participants) | 8
Participants | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to end of study (up to 6.6 years)
Description: Safety Analysis Set included all participants who were enrolled in this Extension Study and who received at least one dose of study medication.
Arm/Group | HYQVIA/HyQvia
All-Cause Mortality (participants affected / at risk) | 1/85
Serious Adverse Events (participants affected / at risk) | 20/85
Other Adverse Events (participants affected / at risk) | 63/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HYQVIA/HyQvia (N=85)
Abdominal pain (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 1
Cardiac failure (Cardiac disorders) | 1
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Conus medullaris syndrome (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papilloedema (Eye disorders) | 1
Pulmonary tuberculoma (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Skin infection (Infections and infestations) | 1
Syncope (Nervous system disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1
Tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Vaginal polyp (Reproductive system and breast disorders) | 1
Ventricular fibrillation (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HYQVIA/HyQvia (N=85)
Abdominal pain (Gastrointestinal disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 6
COVID-19 (Infections and infestations) | 18
Diarrhoea (Gastrointestinal disorders) | 11
Erythema (Skin and subcutaneous tissue disorders) | 5
Fall (Injury, poisoning and procedural complications) | 5
Fatigue (General disorders) | 12
Headache (Nervous system disorders) | 23
Hypertension (Vascular disorders) | 8
Influenza (Infections and infestations) | 8
Infusion site erythema (General disorders) | 13
Infusion site pain (General disorders) | 5
Infusion site pruritus (General disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nausea (Gastrointestinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Pyrexia (General disorders) | 17
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 7
Vomiting (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02955355/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT02955355/SAP_001.pdf